CLINICAL TRIAL: NCT00547014
Title: Oral Administration Of CPG 52364 In Healthy Subjects: A Phase 1, Within-Cohort Randomized, Double-Blinded, Placebo-Controlled, Ascending Single-Dose, Single-Center Study
Brief Title: First Safety Study in Humans of a Single Dose of CPG 52364
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: B1221001; 52364-002
Record Dates: First submitted 2007-10-18; First posted 2007-10-19 (Estimated); Last update posted 2009-03-19 (Estimated); Status verified 2009-03

CONDITIONS: Healthy Volunteers
Keywords: treatment, parallel assignment, double blind, randomized, placebo control, safety study,SLE (Systemic Lupus Erythematosus)
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 1mg (Experimental)
  Interventions: Drug: Placebo Comparator: Cohort 1 Placebo; Drug: 52364 1 mg
- Cohort 2 (Experimental)
  Interventions: Drug: 52364 3 mg; Drug: Placebo Comparator: Cohorts 2, 3, 4 & 5 Two subjects each arm will be assigned to receive placebo
- Cohort 3 (Experimental)
  Interventions: Drug: 52364 10 mg
- Cohort 4 (Experimental)
  Interventions: Drug: 52364 30 mg
- Cohort 5 (Experimental)
  Interventions: Drug: 52364 100 mg

INTERVENTIONS:
Drug: Placebo Comparator: Cohort 1 Placebo — Drug: placebo for cohort 1 as single dose
  Arms: Cohort 1 1mg
Drug: 52364 3 mg — 3 mg capsule single dose administered orally as a single dose
  Arms: Cohort 2
Drug: Placebo Comparator: Cohorts 2, 3, 4 & 5 Two subjects each arm will be assigned to receive placebo — Drug: Placebo for cohorts 2, 3, 4 and 5 administered as a single dose
  Arms: Cohort 2
Drug: 52364 10 mg — Drug: 52364 30 mg capsule as a single dose
  Arms: Cohort 3
Drug: 52364 30 mg — Drug: 52364 30 mg capsule administered as a single dose
  Arms: Cohort 4
Drug: 52364 100 mg — Drug 52364 100 mg capsule administered as a single dose
  Arms: Cohort 5
Drug: 52364 1 mg — 1 mg powder diluted in liquid or placebo (liquid alone) administered orally as a single dose
  Arms: Cohort 1 1mg

SUMMARY:
Determine the safety and tolerability of the study drug, CPG 52364, when given as liquid or capsule. Another purpose is to determine how the drug enters and leaves the blood stream and body tissues over time.

ELIGIBILITY:
Inclusion Criteria:

* Normal body mass index and weight
* No significant diseases in the medical history or clinically significant findings on physical exam, opthalmologic exam, clinical laboratory evaluations or 12-lead electrocardiogram

Exclusion Criteria:

* Current illness or history of medical condition affecting the body's function
* Use of any medication within 7 days, any immunosuppressive medication within 6 months, any investigational drug within 30 days or any vaccine or immunoglobulin within 90 days
* Use of any medications during the study
* Positive TB test
* Smoking within 6 months
* Pregnancy or risk of Pregnancy
* Alcohol or drug misuse within 60 days
* Sensitivity to quinazolines

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2007-09; Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Clinical Assessment of Adverse Events | 28 days/subject

SECONDARY OUTCOMES:
Pharmacokinetic Parameters | 28 days/subject

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1221001&StudyName=First%20Safety%20Study%20in%20Humans%20of%20a%20Single%20Dose%20of%20CPG%2052364